CLINICAL TRIAL: NCT03254173
Title: Mirtazapine for Treatment of Cancer Associated Anorexia-cachexia : a Randomized Controlled Clinical Trial
Brief Title: Mirtazapine for Treatment of Cancer Associated Anorexia-cachexia
Acronym: MCACS100
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Catherine Naseef Hunter (Other)
Responsible Party: Sponsor-Investigator, Catherine Naseef Hunter, Assisstant Lecturer at clinical oncology department at Kasr Al Ainy NEMROCK, Kasr El Aini Hospital
Organization: Kasr El Aini Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MCACS100
Record Dates: First submitted 2017-06-11; First posted 2017-08-18 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Advanced Cancer; Cancer Associated Anorexia - Cachexia
Keywords: Mirtazapine; Anorexia - Cachexia; Advanced Cancer; Appetite
MeSH Terms: interventions — Mirtazapine

STUDY DESIGN:
Intervention Model Description: double-blinded randomized controlled trial.
Who Masked: Participant, Care Provider, Investigator
Masking Description: * Treatment allocation will be concealed from patients, investigators, and study coordinators enrolling the participants.
  * The pills used in the study ( either remeron or placebo ) will be kept into opaque containers , in order to be concealed from patients , investigators and study coordinators.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Active Comparator): Mirtazapine 30 mg oral tablets ( Remeron 30 mg oral tablets ) , as half tablet daily , i.e , 15mg daily , before sleep for a duration of 8 weeks
  Interventions: Drug: Mirtazapine 30 mg oral tablets
- Arm B (Placebo Comparator): Placebo oral tablets , as half tablet daily before sleep for a duration of 8 weeks
  Interventions: Drug: Placebo oral tablets

INTERVENTIONS:
Drug: Mirtazapine 30 mg oral tablets — Mirtazapine 30 mg oral tablets ( Remeron 30 mg oral tablets) , half tablet before sleep for 8 weeks
  Other Names: Remeron 30 mg oral tablets
  Arms: Arm A
Drug: Placebo oral tablets — Placebo oral tablets , half tablet daily before sleep for 8 weeks
  Arms: Arm B

SUMMARY:
A randomized controlled clinical trial will be conducted to assess the efficacy of the FDA approved drug , mirtazapine , in treatment of cancer associated anorexia cachexia syndrome.

Two arms will be compared . Arm A will involve 50 patients with confirmed advanced cancer receiving mirtazapine 15 mg once daily for 8 weeks & Arm B will involve another 50 patients with confirmed advanced cancer receiving placebo for 8 weeks.

Both arms will be compared to assess efficacy of mirtazapine in appetite stimulation primarily and to assess other outcomes secondarily which will be discussed later in details.

DETAILED DESCRIPTION:
* A Written consent is to be obtained from all patients before being enrolled in the study.
* Baseline Complete Blood Count , Liver function tests and kidney function tests will be obtained to assess safety to start the drug and to assess its dose adjustment.
* Two arms will be compared : mirtazapine oral 15mg daily versus placebo. This will be conducted on a double-blinded basis.
* Oral mirtazapine ( REMERON , RD , 30 mg tablets , Organon ) will be the original FDA approved drugs that will be used in the study.
* Treatment allocation will be concealed from patients, investigators, and study coordinators enrolling the participants.
* All patients will be counseled and given dietary advice by a dietician at baseline.
* Patients will be permitted to continue treatment at the same dose as scheduled as long as weight was stabilized (no loss greater than 10 % of body weight at baseline).
* Duration of therapy : Patients will remain on protocol for a duration of 8 weeks as long as they did not develop serious concurrent illness preventing further treatment, unacceptable adverse events (grade 3 or higher), the patient decides to withdraw from study, or the investigator judges that it is in the patient's best interest to discontinue treatment due to general or specific health conditions.
* Demographic data will include performance status, tumor type, sex, age, and percentage weight loss.
* The ESAS scale (Edmonton Symptom Assessment Scale ) will be used to assess the following 10 symptoms experienced by patients with cancer during the previous 24 hours:

  1. pain.
  2. Fatigue.
  3. Nausea.
  4. Depression.
  5. Anxiety.
  6. Drowsiness.
  7. Dyspnea.
  8. Anorexia.
  9. Sleep disturbance.
  10. And feelings of well-being.

The severity of each symptom is rated on a numerical scale of 0 to 10 (0_no symptom, 10_worst possible severity). The ESAS is both valid and reliable in the assessment of the intensity of symptoms in patients with cancer.

* The FAACT questionnaire ( Functional Assessment of Anorexia\Cachexia Therapy ) with anorexia \ cachexia subscale will be used to assess quality of life among the studied patients , in a form of questionnaire including :

  1. Physical well-being.
  2. Social well-being.
  3. Emotional well-being.
  4. Functional well-being.
  5. Additional concerns.

     The patient rates the answer on a scale of 0 to 4. The FACIT - Pal scale is internally consistent , reliable and valid as a measure of health-related quality of life for persons with advanced cancer.

     We will contact their website to get the licence to use the questionnaire and to get its translated version.
* Anthropometric measures to assess efficacy of mirtazapine in weight gain :

  1. Assessment of weight of the patient .
  2. Assessment of muscle strength ( via hand grip dynamometry , using the device named Lite 200 lb , Fabrication Enterprises Incorporated Company).
  3. Assessment of lean ( via bioimpedance analysis , using the device named BF100 , Beurer Company ).
* Biological methods to assess efficacy of mirtazapine in modulating inflammatory cytokine media : quantitative c-reactive protein (CRP) and comparative analysis by enzyme-linked immunoassay (ELISA) will be performed on IL-6 ( Interleukin - 6 ) , and YKL-40 serum levels according to availability. They will be obtained at baseline (day 1 of treatment, immediately before first dose) and at week 8.
* Evaluation of safety and tolerability Patients who will receive at least one dose of study medication will be done.
* A traditional definition of dose-limiting toxicity (DLT) within the first cycle Will be used (any grade 3 non-hematologic or grade 4 hematologic toxicity within 4 weeks and assessed as being at least possibly related to study drug).
* A toxicity questionnaire will be done at baseline and then at 14-day intervals until day 28.

To fully assess the toxicity profile of the drug, the safety evaluation period in the trial will be extended 30 days from the date of the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed advanced cancer.
* Patients with appetite score equal or more than 4 on a 0 to 10 scale (10 _ worst appetite).
* Patients with weight loss more than 5 % of body weight over 6 months . Or : Patients with any degree of weight loss more than 2 % associated with BMI ( body mass index ) of less than 20.
* Patients able to take pills orally and not dependent on tube feeding (no oral mucosal inflammation interfering with oral intake or dysphagia as determined by clinical examination).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* Normal organ function (creatinine ≤2× upper limit of normal, bilirubin ≤2; upper limit of normal).
* Ability to understand and willingness to sign written informed consent.
* Patients could be receiving concurrent chemotherapy or radiation therapy.
* Patients with an expected life span of at least 3 months.

Exclusion Criteria:

* Patients with weight gain for known cause , e.g. , ascites.
* Premenopausal women with childbearing potential with a positive pregnancy test.
* Patients unable to maintain oral intake .
* Patients with dementia or delirium.
* Patients with uncontrolled symptoms that could impact appetite or caloric intake such as nausea, pain, or depression will be excluded until their symptoms had stabilized for at least 2 weeks.
* Because improvement in anorexia and/or weight in depressed individuals could be due to an antidepressant effect of mirtazapine, rather than to a direct effect on anorexia, patients with moderate to severe depressive symptoms will be also excluded. the screening instrument will be a single-item interview assessing depressed mood of the Schedule for Affective Disorders and Schizophrenia (SADS) instrument which is validated and highly accurate in screening for depression when compared to the gold standard of semistructured diagnostic interviews, and is rated on a 6-point Likert scale, where 0 = no depression and 6 = extreme feelings of depression. Patients with a score of 4 or more will be excluded from the study as they are considered to be at high risk for depression.
* No treatment with antipsychotic agents such as risperidone, quetiapine, clozapine, phenothiazine, or butyrophenone for 30 days prior to or during protocol therapy.
* Patients with untreated vitamin B12 deficiency or endocrine abnormalities that could affect appetite, such as thyroid dysfunction and hypoadrenalism.
* Patients on supplements or medications with potential appetite-stimulating activity, such as megestrol acetate, corticosteroids, or thalidomide, will be excluded unless they are put on a stable dose for more than 2 weeks and continue to experience poor appetite.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-03-26 (Actual); Primary Completion 2019-10-17 (Actual); Study Completion 2019-10-17 (Actual)

PRIMARY OUTCOMES:
Efficacy of mirtazapine in appetite stimulation in patients with cachexia due to advanced cancer with a change of increase of 1.5 degree on a numerical scale of 0 -10 as a target . | It will be assessed at week 4 of receiving the intervention. The 4-week duration of treatment is of sufficient length to obtain benefit from an effective intervention for appetite.
  Efficacy of mirtazapine in appetite stimulation in patients with cachexia due to advanced cancer with a change of increase 1.5 degree on a scale of 0-10 as a target , where 0 represents minimum appetite and 10 represents maximum appetite.

SECONDARY OUTCOMES:
Efficacy of mirtazapine in weight gain. ''Improved'' weight will be defined as a gain of ≥ 1 kg and ''maintained weight'' will be defined as a loss of <500 g, or a gain of <1 kg. | It will be assessed at week 8 of receiving the intervention.
  Efficacy of mirtazapine in weight gain in patients with cachexia due to advanced cancer.''Improved'' weight will be defined as a gain of ≥ 1 kg and ''maintained'' will be defined as a loss of <500 g, or a gain of <1 kg.
Effect of mirtazapine in improving other symptoms , such as : nausea , vomiting , sleep with a change of decrease of ≥ 2 points on the ESAS ( Edmonton Symptom Assessment Scale ) from baseline. | It will be assessed at week 8 of receiving the intervention.
  Effect of mirtazapine in improving other symptoms , such as : nausea , vomiting , sleep in patients with cachexia due to advanced cancer with a change of decrease of ≥ 2 points on the ESAS scale from baseline. The ESAS is both valid and reliable in the assessment of the intensity of symptoms in patients with cancer.
Effect of mirtazapine in improving quality of life : will be measured by an increase of 16 points in the FAACT questionnaire ( Functional Assessment of Anorexia\Cachexia Therapy ) with anorexia \ cachexia subscale . | It will be assessed at week 8 of receiving the intervention.
  Effect of mirtazapine in improving quality of life in patients with cachexia due to advanced cancer. This will be measured by an increase of 16 points in the FAACT which indicates ''improved'' quality of life. The FAACT questionnaire ( Functional Assessment of Anorexia\Cachexia Therapy ) with anorexia \ cachexia subscale is internally consistent , reliable and valid as a measure of health-related quality of life for persons with advanced cancer.
  We will contact their website to get the licence to use the questionnaire and to get its translated version.
Changes in inflammatory cytokines associated with mirtazapine administration : quantitative c-reactive protein (CRP) , IL-6, and YKL-40 serum levels . | It will be assessed at week 8 of receiving the intervention.
  Changes in inflammatory cytokines associated with mirtazapine administration in patients with cachexia due to advanced cancer : quantitative c-reactive protein (CRP) and comparative analysis by enzyme-linked immunoassay (ELISA) will be performed on IL-6, and YKL-40 serum levels according to availability. They will be obtained at baseline (day 1 of treatment, immediately before first dose) and at week 8.
Safety of mirtazapine use : Toxicity will be graded according to the Common Terminology Criteria for Adverse Events (CTCAE), version 4.0 | It will be assessed at baseline , then at 14-day intervals until day 28 and after 30 days from the date of the last dose of the study drug.
  Safety of mirtazapine use in patients with cachexia due to advanced cancer.Toxicity will be graded according to the Common Terminology Criteria for Adverse Events (CTCAE), version 4.0. A traditional definition of dose-limiting toxicity (DLT) within the first cycle will be used (any grade 3 non-hematologic or grade 4 hematologic toxicity within 4 weeks and assessed as being at least possibly related to study drug).
  A toxicity questionnaire will be done at baseline and then at 14-day intervals until day 28.
  To fully assess the toxicity profile of the drug, the safety evaluation period in the trial will be extended 30 days from the date of the last dose of study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine N Hunter, Ass. lecturer, Principal Investigator — Clinical Oncology Department at Kasr Al Ainy NEMROCK
Locations (1):
- Kasr Al Ainy - Cairo University - Faculty of Medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All data will be kept in records at clinical oncology department at Kasr Al Ainy NEMROCK to be available at anytime and shared with other researchers